CLINICAL TRIAL: NCT02913937
Title: Comparison of Postoperative Pain and Healing After Passive Ultrasonic Irrigation and Needle Irrigation in Patients With Apical Periodontitis: A Randomized Clinical Trial
Brief Title: Effect of Passive Ultrasonic Irrigation Versus Needle Irrigation on Postoperative Pain and Periapical Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Tawfik aly, postgraduate student, Department of Endodontics, Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-201
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-10

CONDITIONS: Apical Periodontitis
Keywords: ultrasonic irrigation; pain; healing; apical periodontitis
MeSH Terms: conditions — Periapical Periodontitis; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needle irrigation (Active Comparator): Endodontic irrigation will be done using an endodontic needle.
  Interventions: Device: Endodontic needle
- Passive ultrasonic irrigation (Experimental): Endodontic passive ultrasonic irrigation will be done using an endodontic needle followed by passive ultrasonic agitation.
  Interventions: Device: Passive ultrasonic irrigation

INTERVENTIONS:
Device: Passive ultrasonic irrigation — Endodontic irrigation followed by passive ultrasonic agitation.
  Arms: Passive ultrasonic irrigation
Device: Endodontic needle — Endodontic irrigation
  Arms: Needle irrigation

SUMMARY:
The aim of this study is to compare the effect of passive ultrasonic irrigation versus needle irrigation on post-operative pain and healing in patients with permanent posterior teeth with apical periodontitis treated in a single visit.

DETAILED DESCRIPTION:
Full medical and dental history using a dental chart for all patients treated in this study.

Clinical and radiographic examination will be done for all patients to verify the diagnosis of apical periodontitis with periapical radiolucency at least 2mm in diameter.

The treatment protocol and its associated risks and benefits will be explained to the eligible patients before obtaining informed consent. Endodontic procedures will be done in a single visit as follows: access cavity preparation using sterile round bur and Endo-Z bur, isolation using a rubber dam, canal preparation using a nickel-titanium rotary system then obturation. During mechanical preparation, irrigation will be done using passive ultrasonic irrigation (Experimental group) where ultrasonic activation will be done for irrigant-filled canals using the U- file tip (Varios NSK) in an ultrasonic device (P5 Newtron; Satelec Acteon) 1mm from the working length after each file change for 10 sec, or needle irrigation (Control group) where only the endodontic irrigation needle will be used; the irrigation protocol for each patient will be determined following a random-number sequence.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-55 years old.
* Males and females.
* Positive patient's acceptance to participate in the study.
* Mature, permanent, mandibular, posterior teeth with apical periodontitis.

Exclusion Criteria:

* Medically compromised patients so that no other pain source or drug interaction could interfere with pain resulting from the endodontic therapy.
* Patients who had received analgesic treatment recently (past 8 hours) as it can affect the results
* Pregnant females.
* Teeth with previous root canal treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 7 days
  postoperative pain will be assessed using numerical rate scale (NRS).

SECONDARY OUTCOMES:
Periapical healing | 12 months
  Periapical healing will be assessed using periapical index (PAI).

CONTACTS AND LOCATIONS:
Overall Officials: Randa El-Bogdady, Study Director — Cairo University; Suzan AW Amin, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gondim E Jr, Setzer FC, Dos Carmo CB, Kim S. Postoperative pain after the application of two different irrigation devices in a prospective randomized clinical trial. J Endod. 2010 Aug;36(8):1295-301. doi: 10.1016/j.joen.2010.04.012. Epub 2010 Jun 19. PMID 20647083
- [Background] Middha M, Sangwan P, Tewari S, Duhan J. Effect of continuous ultrasonic irrigation on postoperative pain in mandibular molars with nonvital pulps: a randomized clinical trial. Int Endod J. 2017 Jun;50(6):522-530. doi: 10.1111/iej.12666. Epub 2016 Jun 28. PMID 27248848